CLINICAL TRIAL: NCT06768294
Title: Baricitinib in Calcium PyrophosphAte DePosiTion DIseaSe Trial - a Proof of Concept Phase II Clinical Trial
Brief Title: Baricitinib in CPPD - the BAPTIST Study
Acronym: BAPTIST
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Baptist (L4194)
Record Dates: First submitted 2024-11-04; First posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Calcium Pyrophosphate Deposition Disease; Chondrocalcinosis
Keywords: calcium pyrophosphate deposition disease; chondrocalcinosis; pseudogout; ultrasound; baricitinib; olumiant; synovial biopsy; arthritis
MeSH Terms: conditions — Chondrocalcinosis; Arthritis | interventions — baricitinib; Methylprednisolone; Adrenal Cortex Hormones; Colchicine; Hydroxychloroquine; Methotrexate; Folic Acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- One group will receive baricitinib at the dose of 4mg/daily (Active Comparator)
  Interventions: Drug: Baricitinib 4 MG Oral Tablet
- standard of care (to be decided according to the guidelines) (Sham Comparator): Methylprednisolone tablets, Colchicine 1 mg tablets, Hydroxychloroquine 200 mg tablets, MTX + folic acid (to be decided according to the guidelines)
  Interventions: Drug: Methylprednisolone (Corticosteroid); Drug: Colchicine 1 MG Oral Tablet; Drug: Hydroxychloroquine 200 mg; Combination Product: Methotrexate + Folic Acid

INTERVENTIONS:
Drug: Baricitinib 4 MG Oral Tablet — Baricitinib is a JAK1/JAK2 inhibitor approved for use in Rheumatoid Arthritis. It is under investigation for use in several inflammatory diseases, including Psoriasis and Psoriatic Arthritis, Atopic Dermatitis, Inflammatory Bowel Disease and Systemic Lupus Erythematosus, with encouraging results. As IL-6 plays a central role in CPPD inflammatory process, a broad spectrum of interleukins and other proinflammatory proteins (including interferons) could be involved. A drug that acts by blocking more than one proinflammatory cytokine could be a promising treatment for a multifaceted disease such as CPPD.
  Arms: One group will receive baricitinib at the dose of 4mg/daily
Drug: Methylprednisolone (Corticosteroid) — The initial dosage of methylprednisolone may vary depending on the entity of inflammation and the patient's comorbidities. Usually in CPPD a short-term administration of methylprednisolone starts with 16 mg per day after breakfast decreasing the initial dosage in small decrements at appropriate time intervals until discontinuation, in about 2 weeks. Methylprednisolone will be given in combination with gastroprotective agents such as proton pump inhibitors.
  Arms: standard of care (to be decided according to the guidelines)
Drug: Colchicine 1 MG Oral Tablet — 1 or ½ tablet (depending on individual tolerance) daily after breakfast
  Arms: standard of care (to be decided according to the guidelines)
Drug: Hydroxychloroquine 200 mg — 1 tablet daily after lunch
  Arms: standard of care (to be decided according to the guidelines)
Combination Product: Methotrexate + Folic Acid — MTX 2.5 mg tablets, from 2 to 4 tablets (5-10mg), depending on disease severity, to be administered once weekly after dinner, always in the same day of the week. One tablet of folic acid (folina 5 mg) will be administered the day after MTX administration, after breakfast, to reduce and prevent the common side effects of MTX.
  Arms: standard of care (to be decided according to the guidelines)

SUMMARY:
The aim of this clinical trial is to determine if baricitinib is effective in treating calcium pyrophosphate deposition disease (CPPD) in adults. The primary objective is to assess its impact on joint inflammation. The key questions the study seeks to answer are:

* Can baricitinib reduce inflammation in affected joints?
* Will baricitinib lead to changes in ultrasound findings, such as calcium crystal deposition and synovitis?

Researchers will compare baricitinib to other treatments, including methylprednisolone, colchicine, hydroxychloroquine, and methotrexate with folic acid, for managing CPPD.

DETAILED DESCRIPTION:
Calcium Pyrophosphate Deposition disease (CPPD) is a frequent arthropathy in the elderly (over 55 years old), varying from 7% to over 45% depending on the diagnostic method used (X-rays, ultrasonography, synovial fluid analysis, or microscopic analysis of tissues) and the age of the sample group. No data are available on the incidence of the disease. Osteoarthritis (OA) and CPPD are usually associated (aging is a common risk factor for both diseases), but their relationship is not clear even if CPPD is believed to be a primary factor that causes joint damage and worsens the clinical outcome of OA. Recent evidence highlights substantial differences between the two diseases with OA and concomitant CPPD presenting a higher degree of inflammation in both the monoarticular and polyarticular phenotype, resembling more a seronegative arthritis than a prevalent degenerative disease alone. Increasing interest in CPPD is underlined by the recent proposal for a creation of a specific Outcome Measures in Rheumatology (OMERACT) group aimed at establishing the core domains of the disease and the proper instruments for disease diagnosis and assessment over time. Currently, no specific treatment for this disease has been identified. The first line of treatment is designed to reduce pain and inflammation using symptomatic drugs (steroids, non-steroidal anti-inflammatory drugs [NSAIDs], colchicine) that demonstrate some efficacy but are unsuitable for long-term use. Other drugs have been tested in spontaneous observational studies (methotrexate [MTX], interleukin-1 [IL-1] inhibitors), though data on their efficacy is controversial. Similarly, anti-tumor necrosis factor (TNF)α drugs also seem to have limited effect on the inflammation in CPPD disease.

The Janus kinase (JAK) family of non-receptor tyrosine kinases transduce signals from multiple cytokines, including IL-6, and growth factors. Baricitinib is a JAK1/JAK2 inhibitor approved for use in Rheumatoid Arthritis. It is under investigation for use in several inflammatory diseases, including Psoriasis and Psoriatic Arthritis, Atopic Dermatitis, Inflammatory Bowel Disease and Systemic Lupus Erythematosus, with encouraging results[4]. As IL-6 plays a central role in CPPD inflammatory process, a broad spectrum of interleukins and other proinflammatory proteins (including interferons) could be involved. A drug that acts by blocking more than one proinflammatory cytokine could be a promising treatment for a multifaceted disease such as CPPD.

At the moment there are no drugs with precise indication for use in CPPD. Published recommendations of the task force of the European League Against Rheumatisms (EULAR), based on the mechanism of action of the drugs used in chronic arthritis, on the scarn literature and on expert's opinion, suggest the use of non-steroidal anti-inflammatory drugs (NSAIDs) and local or systemic steroids for acute attacks combined if necessary with colchicine and the use of hydroxychloroquine or methotrexate for the use in chronic arthritis. Colchicine may also be used for prophylaxis in case of frequent acute attacks of arthritis. A recent European retrospective study on the treatment of CPPD demonstrated that colchicine and methotrexate were the most frequently used first line drugs for chronic CPPD and demonstrated to be efficient (significant improvement) in 41.9% of patients for colchicine and 58.3% for MTX. The 24 months retention rate was 29.1% for colchicine and 44.4% for MTX. Hydroxychloroquine also demonstrated a good efficacy (improvement in 87.5% of patients) but only a small number of patients were in treatment with such drug .

In summary, many features of CPPD are still unclear and need to be investigated. Basic and clinical research is necessary to understand the disease's pathogenetic mechanisms and possibly amplify the efficacy of available treatments. The failure or partial efficacy of drugs that block only one proinflammatory protein indicates that the pathogenesis of the disease involves more than one pathway. We are therefore interested in testing Baricitinib as a potential treatment in CPPD by synovial, clinical, ultrasound and biochemical Study in a pilot study.

All participants will benefit a tight study visit of the disease and their symptoms during the study with accurate monitoring and will be granted the most up-to-date treatment modalities for this disease. The interventional drug, already in commerce and used for patients with Rheumatoid arthritis and other inflammatory conditions (Juvenile inflammatory arthritis, atopic dermatitis) ), has been highly effective in reducing inflammation and joint pain. Further, baricitinib blocks one of the most expressed proinflammatory cytokines in CPPD, IL-6, raising the possibility of improved outcomes in this disease.

Therefore, the study could open the way for phase II and III trials, giving hope to all patients with CPPD for a treatment option, as there is no drug with a specific indication for CPPD.

In the early years of JAK inhibitors (JAKi) in clinical practice, concerns arose about cardiovascular and thromboembolic events, particularly with tofacitinib, prompting a comprehensive evaluation of the entire drug class. However, real-world data have been reassuring. A recent editorial reviewing pre- and post-marketing studies for tofacitinib, baricitinib, and upadacitinib in rheumatoid arthritis, psoriatic arthritis, and axial spondyloarthritis highlights that the actual risk of major cardiovascular events (MACE) in patients with inflammatory diseases remains unclear. Post-marketing studies have shown no significant increase in MACE incidence and, in some cases, a lower incidence in RA patients treated with baricitinib.

The incidence of adverse events (AEs) does not appear to correlate with JAKi dosage but may be linked to high disease activity, as persistent inflammation is a known risk factor for MACE. The analysis suggests that major risk factors for MACE during baricitinib treatment include a history of MACE and advanced age (though no specific threshold is provided). In this study, patients with recent MACE (&lt;6 months) will be excluded. Those with a more distant history of MACE will undergo a thorough cardiovascular risk assessment and may be enrolled based on the clinician&#39;s judgment, considering that persistent joint inflammation is a risk factor for MACE and should be treated. Finally, an important aspect to keep in mind are the recent findings that suggest that acute CPPD arthritis is also a risk factor for MACE.

Therefore, taking under consideration all the above mentioned issues, the increase of cardiovascular risk in patients with uncontrolled inflammation and the possible adverse events in patients with specific risk factors, only patients that have a clearly favourable benefit/risk profile will fulfil both the inclusion and exclusion criteria and could be enrolled in the study.

The primary aim of this proof-of-concept study is to evaluate the effect of baricitinib on inflammation of the synovial membrane in CPPD. The outcome for the primary objective is the changes in the synovial tissue CD68 scoring at 12 weeks, an objective outcome measure.

The secondary objectives of the study are:

* To assess changes in Krenn synovitis score and cytokines at the synovial level;
* To evaluate the improvement of patient-reported outcomes (PROs) and pain;
* To determine changes at ultrasound examination in terms of calcium crystal deposition, synovitis and degenerative changes;
* To identify subsets of the disease that could have a better response to the treatment;
* To evaluate the effect of baricitinib on serum cytokine levels at a plasmatic level.

Finally, exploratory objectives of the study are:

* To explore the possible baricitinib-induced impact on whole-body metabolism;
* To explore differences in biochemical and immunohistological markers between patients with the acute and the chronic form of CPPD.

The result of baricitinib will be tested against the standard of care for CPPD arthropathy as defined by the 2011 recommendations for managing CPPD.

This is a single-centre, National, prospective, monocentric, randomized, controlled, phase II pharmacological trial. Consecutive patients reaching the outpatient clinic of the IRCCS Ospedale Galeazzi - Sant'Ambrogio in an 18-month period satisfying the 2023 American College of Rheumatology (ACR)/EULAR classification criteri for CPPD disease, belonging in any of the clinical subsets of CPPD described below, will be enrolled and randomized in two groups. One group will receive baricitinib at the dose of 4mg/daily, while the second group will receive the standard of care, for a total number of 32 patients, 16 for each group. Randomization and drug administration will be carried out by one operator, while clinical, laboratory and ultrasound assessments and histological examinations will be carried out by different operators blind to patients' treatment arms.

The study include tree different phases:

1. Screening/Enrolment: phase for patients selection and consent collection. Screening and Enrolment may coincide
2. Treatment: phase of drugs administration (Baricitinib or comparator); the treatment period consists of 24 weeks of drug administration, so it coincides with the study visits.
3. Study Visits: 24 weeks of therapy control punctuated by visits at week 4, 12 and 24.

The total expected duration for the clinical study is 28 months, of which:

* From month 0 to month 18 for enrolment
* From month 1 to month 24 for Study Visits The unblinded clinician will provide all drugs at each visit in adequate quantity to reach the next study visit.

Number of tablets of each medication delivered to the patients and the effective number of consumed tablets will be registered at each visit.

All drugs listed in the protocol will be stored, labelled and dispensed to the doctor by the Institute Pharmacy located in the Hospital itself. Any residual medicine will be destroyed at the end of the study by the Pharmacy according to institute procedures. The Pharmacy, certified with adequate quality certification, will follow the internal procedures approved by the Institution for the management of experimental drugs.

The unblinded clinicians and the Pharmacy (see below) will keep a cumulative inventory and dispensing records and will maintain all supplies under adequate security conditions. Adequate record of receipt and use or loss of drug will be retained. This inventory record must be available for inspection by at any time.

For each patient enrolled, complete demographic (age, sex, type of occupational activity, smoking habit) and anthropometric data (height and weight) will be recorded. Furthermore, complete anamnestic data will be collected. Notably, they will include information about previous or current therapies (both continue and on-demand, including steroids, NSAIDs, DMARDs, and biological DMARDs), the date of the symptom onset, the disease duration and the main comorbidities.

All the patients will undergo a physical examination to assess the presence of tender and swollen joints according to the 44 swollen joint counts and Ritchie articular index.

A co-investigator, blind to treatment allocation, ultrasound and laboratory findings, will carry out the clinical examination. The blinding of this investigator will be ensured with patient training and information compartmentalization. Patients will be worn to avoid telling the doctor the drug that he/she is taking. Furthermore, all the personnel involved in the study will be instructed not to reveal to the blinded investigator patients' therapies. This investigator will not have access to the clinical and/or experimental material in which the therapeutic indication is reported and will perform only the clinical examination. Finally, the primary outcome of the study is an objective, quantitative measure and the personnel that will perform the analysis will not have any contact with the patients. This will ensure the blinding for the primary endpoint of the study. During the visits will be recorded any concomitant treatments. All patients will fill in the following PROs independently before the clinical assessment: HAQ, WOMAC and a VAS for pain at the involved joints.

Standard blood exams will include: ESR, hsCRP, blood count, transaminase, creatinine, ferritin, total calcium, ionized calcium, inorganic phosphate, magnesium, 25(OH)vitamin-D, intact PTH, total cholesterol, LDL, HDL, triglycerides, CPK. Circulating cytokines dosage will include IL-1, IL-6, IL-8, anti-TNFα, Interferon α and γ, and TGFβ.

The ultrasound assessment will include the wrists and hands, knees and the affected joints if different than hands/wrists/knees. It will be performed at baseline, 4, 12 and 24 weeks. The ultrasound elementary lesions and the scores will be provided following the published definitions. Ultrasound examinations will be carried out by an operator blind to the treatment and to clinical/laboratory findings according to the EULAR standardised procedures for ultrasound.

Synovial tissue will be obtained by US-guided biopsy of an affected joint at baseline (enrolment) and from the same joint 12 weeks after treatment. The biopsy procedures will be carried out in a clean procedure room. Ultrasound biopsy procedure follows a similar routine with 1-3 mL of local anaesthetic (1% lidocaine) injected into the soft tissues up to the joint capsule, visualized under US guidance. A further 2-5 mL of local anaesthetic (1% lignocaine) will be instilled into small joints, 10-15 mL for large joints. For larger joints, a suitable coaxial outer needle may be used in addition to the Core Biopsy Needle (from 14G to 18G, depending on the site) placed within the joint capsule. A longitudinal US image will be used to detect the needle and guide it to an appropriate predetermined site for biopsy. For smaller joints, a Quick-Core biopsy Needle (16G, throw length 10 mm) will be used without a coaxial sheath. The maximum tolerated number of biopsies per joint will be attempted with the aim for a minimum of 8-12 biopsies to be retrieved per procedure. Following the procedure, a small sterile dressing will be placed over the needle insertion site. Typically, this procedure will last from 30 to 45 min from the instillation of anaesthetic to the final biopsy. There is little difference in the duration of procedures from small to large joints.

Histological analyses of the synovial tissue will be performed at the Laboratory of Experimental Biochemistry of IRCCS Istituto Galeazzi-Sant'Ambrogio, Milan (Italy).

An operator will carry out a synovial tissue examination, blind to treatment allocation, clinical, laboratory and ultrasound findings.

The chronic inflammation may favour metabolic homeostasis towards oxidative and low energy availability.

Targeted metabolomics analysis will be performed on blood samples (baseline, 12 and 24 weeks) to quantify the changes in the energy metabolism molecules. Parallel untargeted metabolomics analysis on the same samples will be performed using standardized bioinformatics tools to discover the most relevant metabolic pathways involved in the pathogenesis of CPPD and/or valuable to monitor the therapeutic path of the CPPD patient.

Targeted metabolomics will be done to quantify key small molecules involved in the energy cycles and oxidative stress. In this analysis, the metabolites will be extracted from the serum and then their concentrations will be compared to the analytical standards.

Untargeted metabolomics will be performed to profile the whole small molecule composition in the serum of enrolled patients compared with the standard non-treated healthy individuals. In this analysis, metabolites will be extracted from samples and analysed using high-resolution liquid mass spectrometry. Results will generate the complete profile of metabolites and small molecules in the serum of patients compared to standardized samples. Using different bioinformatics tools then, it will be possible to create a functional network of crucial metabolites and possibly the active enzymes involved in the procedure.

The data generated in this study will be recorded at the study site by the appointed study personnel on a study-specific, validated (as per 21 CFR Part 11 requirements) electronic Case Report Form (eCRF). eCRFs will be designed in order to act as a reminder both as far as the timing and the nature of the data to be collected are concerned. The initial (entry) page will specify how to fill them in, in agreement with satisfactory regulatory standards.

eCRFs will be designed by the appointed eCRF Designer of the CRO's Data Management Unit, using a validated clinical data management system.

In agreement with satisfactory regulatory standards, the investigators, study coordinators, and study monitors will be instructed on the proper use of the electronic eCRF system and provided with a user manual with appropriate instructions on software usage, together with individual, private User ID and Password to have access to the eCRF. The name of personnel authorized to complete an eCRFs are to be given to the assigned study monitor before trial initiation. Data entered in the eCRF will be captured by a fully validated system and stored in a dedicated electronic database at the CRO site, properly designed by the Data Manager, which will be used to produce all planned statistical analyses. All patient data will be reported on the eCRF in a pseudo-anonymous fashion, identifying the patient only through a patient number.

The Investigator will be responsible for the completeness, accuracy and timeliness of the data reported. All source documents should be completed in a neat, legible manner to ensure the accurate interpretation of data. The Investigator is required to verify the data transcribed onto the eCRFs.

The eCRF should be filled-in during or immediately after the conclusion of each visit, preferably within 24 hours but no later than five working days after the visit.

The study monitors then have to check the eCRFs against the source documents for accuracy and validity, as applicable. All clinical data recorded on the eCRF will be coded and identification is restricted to authorized personnel involved in the study and under the responsibility of the researcher. It is possible that the clinical data of the subject are stored and processed electronically for purposes of scientific evaluation, but any discussion or analysis of the data will always be done anonymously. Clinical, laboratory and ultrasound data will be collected by Investigator, or designated member of the Investigator's staff, into the clinical case report forms prepared ad hoc for this study, and then inserted in an eCRF by the data manager, in order to maintain blinding between investigators. A unique ID composed by the identification code of each investigator will be created (the first two letters of name and surname).

Patients will be registered on study eCRF; the name of the patient will not be recorded. A sequential identification number will be automatically attributed to each patient registered in the trial. This number will identify and must be included on all CRFs, scale, questionnaire and other trial related documents or communications. Explicit consent for the processing of personal data will be obtained from the participating subject (or his/her legally acceptable representative) before collection of data. As anticipated above, computer systems used for remote data collection and the system for data storing and processing are validated. Verification and cross-verification of the data entered by the study personnel at each visit will be automatically performed by the system, according to predefined nature/type of the data, value ranges and rules. All rules applied by the system to check specific items will be detailed in a document issued by the Data Management service of the CRO. Queries will be automatically generated by the system for all data found to be inconsistent, incorrect or missing. Queries to be solved/unclear data to be corrected (or confirmed) will be highlighted by the system, to be easily identified by the study personnel when accessing the eCRF website. All changes performed by the Investigator will be tracked by the system. During the study, the monitoring will be prevalently made by e-mail and telephone. A data review will be done (by the data manager), at least once a month, mainly to check data inconsistencies, the completeness of patient records, the adherence to the protocol and to Good Clinical Practice and the progress of enrolment. Once all data have been entered in the eCRF and all outstanding queries have been solved, the Monitor of the study will authorize the Investigator to "freeze" the data of the patient's eCRF. No change will be accepted by the system after freezing. Nonetheless, it may be still necessary to edit additional queries following general quality control checks performed by the Data Manager of the study on the frozen.

database: in case, queries will be edited in paper form and referred to the appropriate hospital/study site personnel, to be resolved with assistance of the study Monitors.

When all data are received, all data problems have been resolved, all data checks and quality control checks have been performed, and a blind data review meeting has been held, the trial database is considered clean and can be locked. Any changes to the database after that time can only be made by joint agreement between the Clinical Study Manager, the Statistician, and the Data Manager.

After database lock, the planned statistical analysis will be performed. Any further modification of recorded data will be documented in a database log form.

All Adverse Events (AEs) will be recorded in the eCRF constantly throughout the trial.

Descriptive statistics will be provided in summary tables according to the type of variable. Continuous variables will be summarized by descriptive statistics (number of cases, mean, standard deviation (SD), median, first and third quartile, minimum and maximum). Categorical variables will be summarized using counts of patients and percentages.

Before being included in the study, patients who meet all the criteria for inclusion and exclusion of the study, should be informed in detail by persons delegated by the principal investigator and be placed in a position to understand the objective, meaning, and duration of the study. All the risks/benefits, advantages/disadvantages must be discussed with the subject.

In seeking informed consent, the Investigator will inform the patient that participation to the study is voluntary and that refusal will not lead to loss of any benefit or prejudice the relationship with the physician in any way. Furthermore, a statement will be made to the effect that withdrawal from the study is possible at any moment without having to give a specific reason.

Before admission to the study, the subject must give their written informed consent by signing and dating the form, of which they will receive a signed copy. The subject is guaranteed that participation in the study is voluntary and that at any moment they can withdraw from the study without suffering any consequences.

The researcher conforms to the principle of the right of the subject to the protection of privacy under Legislative Decree no. 196/2003 and ssm, UE Regulation 679/2016 and Guidelines of the Data Protection Authority of 24/07/2008.

To protect the patient&#39;s identity, the Investigator will assign each patient a patient identification code to be used instead of the patient&#39;s name when reporting adverse events or other trial related data. Personal information will be confidential, but may need to be reviewed by authorised representatives and regulatory authorities. Consent to allow direct access to original medical records for data verification purposes must be obtained from the patient prior to participation in the study.

All clinical data recorded on the eCRF or used for further evaluation are coded by number of patient, date of birth and identification is restricted to authorized personnel involved in the study and under the responsibility of the researcher. Clinical data of the subject will be stored and processed electronically for purposes of scientific evaluation, but any discussion or analysis of the data will always be done anonymously.

Results from the medical examinations, instrumental and laboratory tests will be recorded in the patient eCRF. All the information obtained during the conduct of the study with regard to the patient&#39;s state of health will be regarded as confidential and agreement must be obtained prior to the disclosure of his/her personal identity to a third party different from authorised personnel of the study Sponsor and/or Competent Authority.

It is possible that the clinical data of the subject are stored and processed electronically for purposes of scientific evaluation, but any discussion or analysis of the data will always be done anonymously.

IRCCS Ospedale Galeazzi-Sant'Ambrogio (Milan, Italy) owns all data collected in the course of this trial. Investigators and Institutions involved in the clinical trial will enable monitoring, audits and regulatory inspections related to the clinical trial. This include providing direct access to original data and documents.

The Principal Investigator accepts herewith to treat any unpublished information as confidential and ensures that confidentiality is kept also by all staff involved in this project. The investigator should inform the patient&#39;s General Practitioner of the patient&#39;s participation in the trial, if the patient agrees.

In case of a breach of data confidentiality, the Principal Investigator will inform the Institute Data Protection Officer to evaluate possible strategies aimed at limiting the resulting damage.

A clinical study report (CSR) will be prepared according to ICH topic E3 guidelines. An interim and a final CSR will be prepared once the results of the interim and the final analysis will be made available, respectively.

The report will include a thorough description of the relevant methods, a discussion of the results, and a list of all the measurements.

A draft of the CSR will be submitted to the Principal Investigator for comments. After receiving the comments, or two months later if no comments are received, a final version of the CSR will be issued. Any subsequent modification will be considered as an amendment to the CSR. The Investigator's agreement and signature will be obtained. The signed original of the CSR will remain with the study promoter. At the end of the study the IEC and Competent Authority will receive a summary of the CSR.

The preliminary results of this study, as well as the final results, in the form of manuscripts, to be submitted to national and/or international Journals, as well as posters/oral communication at national and/or international Congresses could be reported by the Investigators by IRCCS Ospedale Galeazzi-Sant'Ambrogio authorization.

All investigators participating in this study will be granted authorship for all publications that include collected data. The authors of this protocol will be given authorship for all kinds of publications independently from personal contributions.

Anyway, the publication will neither disclose the identity of patients, fully respecting the data protection laws now in force, nor any patent information.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent;
* Male and female patients aged ≥55 years;
* Patients that according to the investigator's judgement will benefit from the proposed treatments (favourable benefit/risk profile)
* Menopause for women;(no menses for 12 months without an alternative medical cause. A high follicle stimulating hormone level in the postmenopausal range may be used to confirm a postmenopausal state in women not using hormonal contraception or hormonal replacement therapy. However in the absence of 12 months of amenorrhea, a high follicle stimulating single measurement is insufficient.);
* Male patients must avoid having a child during the trial and must use one of the highly effective methods of contraception or sexual abstinence or have a menopause partner (no menses for 12 months without an alternative medical cause. A high follicle stimulating hormone level in the postmenopausal range may be used to confirm a postmenopausal state in women not using hormonal contraception or hormonal replacement therapy. However in the absence of 12 months of amenorrhea, a high follicle stimulating single measurement is insufficient). Contraception methods include:

  * Total abstinence (when this is in line with the preferred and usual lifestyle of the subject). Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
  * Sterilization of the female partner (have had surgical bilateral oophorectomy with or without hysterectomy), total hysterectomy or tubal ligation at least six weeks before the partner enrollment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow-up hormone level assessment
  * Male sterilization (vasectomy) at least 6 months prior to screening
  * Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps).
  * The female partner use oral, (estrogen and progesterone), injected or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS)
* Patients fulfilling the 2023 ACR/EULAR classification criteria for CPPD disease;
* Patients with feasibility of synovial biopsy at the knee or wrist joint;
* Patients with CPPD clinical presentation that may be:

  * Subset 1: patients with prevalent polyarticular involvement of the small joints and tendons of hands and wrists (rheumatoid-like subset). Patients that present with prevalent inflammatory involvement of the hands and wrists (joints and/or tendons), with or without acute attacks of arthritis of the large joints, will be included in this group. Inclusion criteria will be joint effusion and/or synovitis of the II and/or III metacarpal phalangeal (MCP) joint of at least one hand, tenosynovitis of at least 1 tendon of one hand or wrist, hyperostosis of the II and/or III MCP head;
  * Subset 2: patients with prevalent involvement of the large joints (oligoarthritis). Patients with recurrent/persistent effusion in one or more large joints (independently of the presence and grade of OA), not responsive to a single injection of steroid and white cell count in joint synovial fluid that is more than 2000 cells/mm3 and/or patients with acute monoarticular arthritis, with more than 3 attacks in one joint in the last 12 months, will be included in this group.

Exclusion Criteria:

* Patients positive at anticitrullinated positive antibodies (ACPA), any titre;

  * Patients affected by seronegative arthritis or other conditions that may be responsible of arthritis (i.e. gout, rheumatic polymyalgia, etc);
  * Patients that refuse synovial biopsy or present contraindications, according to investigator's judgement, including (but not limited to) increased risk for bleeding (platelet count <100000 or use of anticoagulants), allergy to local anesthetics, suspicion of septic arthritis;
  * Patients with history of malignancy or lymphoproliferative disease; or have signs or symptoms suggestive of possible lymphoproliferative disease, including lymphadenopathy or splenomegaly; or have active primary or recurrent malignant disease; or have been in remission from clinically significant malignancy for < 5 years;
  * Patients with cervical carcinoma in situ, basal cell carcinoma or squamous cell carcinomas who have had active disease within 3 years of screening for this study;
  * Patients with active, untreated, acute or chronic infection (such as untreated tuberculosis), or immunocompromised to an extent that such that participation in the study would pose an unacceptable risk to the subject. Patients with treated infections such as latent tuberculosis after completion of the appropriate therapy are not excluded;
  * Patients with clinically serious infection or that have received intravenous antibiotics for an infection, within 4 weeks of randomization;
  * Patients with active viral infection that, based on the investigator's clinical assessment, makes the patient an unsuitable candidate for the study;
  * Patients with serology suggestive for active or chronic hepatitis B or hepatitis C infection; anti-HCV, anti-HBs, anti-HBc antibodies and HBcAg, HBsAg will be tested. Patients that will result positive for anti-HCV and/or HBcAg and/or HBsAg and/or anti-HBc antibodies will be excluded from the study. Patients who are positive for both anti-HBc and antiHBs, but negative for HBcAg and HBsAb could be enrolled.
  * Patients with symptomatic herpes zoster infection within 12 weeks of screening or recurrent or disseminated (even a single episode) herpes zoster;
  * Patients with a history of disseminated opportunistic infections (e.g., listeriosis and histoplasmosis);
  * Patients with a history of venous thromboembolism (VTE), or are considered at high risk for VTE as deemed by the investigator
  * Patients who are currently on immunosuppressive therapies or have not discontinued them for at least 4 weeks;
  * Patients with clinically significant (per investigator's judgement) drug or alcohol abuse within the last 6 months preceding the baseline visit;
  * Patients with any major surgery within 8 weeks prior to baseline or requiring major surgery during the study, which in the opinion of the investigator would pose an unacceptable risk to the patient;
  * Patients with recent (within past 6 months) cerebrovascular accident, myocardial infarction, coronary stenting and uncontrolled hypertension (confirmed systolic blood pressure >160 mmHg or diastolic blood pressure >100 mm Hg); patients with less recent major cardiovascular events (> 6 months) will be thoroughly assessed for cardiovascular risk taking under consideration all possible risk factors and the disease phenotype and activity and will be included only in case of favourable benefit/risk ratio according to the principal investigators judgement.
  * Patients with presence of significant uncontrolled respiratory, hepatic, renal, endocrine, hematologic, neurologic, or neuropsychiatric disorders, or abnormal laboratory screening values that, in the opinion of the investigator, pose an unacceptable risk to the patient if participating in the study or of interfering with the interpretation of the data;
  * Patients with clinical laboratory test results at screening that are outside the normal reference range of the population and are considered clinically significant, or have any of the following specific abnormalities: neutrophil count <1500 cells/µL, lymphocyte count <500 cells/µL, platelet count <100,000 cells/µL, aspartate transaminase (AST) or alanine aminotransferase (ALT) > 2 times the upper limit of normal, haemoglobin <10 g/dL for male and female subjects, eGFR < 30 mL/min;
  * Patients with any other condition that precludes him/her from following and completing the protocol, in the opinion of the investigator;
  * Patients currently enrolled in or discontinued from a clinical trial involving an investigational product or non-approved use of a drug or device within the last 4 weeks or a period of at least 5 half-lives of the last administration of the drug, whichever is longer, or concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study.
  * Hypersensitivity to the active substance or to any of the excipients

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
The evaluation the effect of baricitinib on inflammation of the synovial membrane in CPPD | The outcome for the primary objective is the changes in the synovial tissue CD68 scoring at 12 weeks, an objective outcome measure.
  CD68 score will be used as outcome measure for the primary objective. CD68 score will be calculated from an analysis of 6 images from each biopsy section and expressed as the mean area of tissue occupied by positively stained cells.

SECONDARY OUTCOMES:
To assess the changes in Krenn synovitis score at the synovial level | 12 weeks
  Krenn score will be used to determine the degree of synovitis according to the three synovial membrane features: synovial lining cell layer, stroma cell density, and inflammatory infiltrate. All parameters will be graded with a semiquantitative score (from 0 to 3) as follows: 0 (absent), 1 (slight), 2 (moderate) and 3 (strongly positive). All parameters will be summarized with a final total score by adding the score of the single features (will range from 0 to 9) and interpreted as follows: 0-1: no synovitis; 2-4: low-grade synovitis; 5-9: high- grade synovitis.
To assess the changes in cytochin levels at the synovial membrane | 12 weeks
  The biopsy samples will be immediately placed in 10% neutral buffered formalin fixed for 48 h and embedded in paraffin for histologic and immunohistochemical analyses. Overall staining intensity will be evaluated. The overall score of the staining intensity will be graded in a four degree scale: negative (0), weak (1), moderate (2), and strong (3).
To determine changes at ultrasound examination in terms of calcium crystal deposition | 4, 12 and 24 weeks
  The ultrasound assessment will include the wrists and hands, knees and the affected joints if different than hands/wrists/knees. For CPP deposition, the CPP deposits of knees, wrists and any involved site will be scored with a semi-quantitive score (0-3).
To determine changes at ultrasound examination in terms of synovitis | 4, 12 and 24 weeks
  The ultrasound assessment will include the wrists, hands, knees and the affected joints if different than hands/wrists/knees. Synovitis will be scored according to the semiquantitative Global OMERACT EULAR Scoring System (GLOESS), a semiquantitative score (0-3) that can be interpreted as: no inflammation (0), slight inflammation (1), moderate inflammation (2) and severe inflammation (3)
To determine changes at ultrasound examination in terms of bone changes | 4, 12 and 24 weeks
  The ultrasound assessment will include the wrists and hands, knees and the affected joints if different than hands/wrists/knees. Bone profile irregularities intended as erosions and/or osteo-proliferative changes (osteophytes) will be scored with a dichotomic score (0: absence, 1:presence).
To evaluate the effect of baricitinib on serum cytokine levels at a plasmatic level. | 12 and 24 weeks
  Blood exams will include circulating cytokines dosage will include IL-1, IL-6, IL-8, anti-TNFα, Interferonα and γ, and TGFβ. For cytokine analysis, blood will be immediately centrifuged at 1300g (10 min, 15°C) and serum will be aliquoted and stored at -80°C until assayed. Cytokine concentrations will be assayed in serum by means of customized high-sensitive magnetic beads-based immunoassays, following manufacturer's protocol. Assays will be performed using a Luminex® MagPix instrument. The sensitivities of the assays are: 0.29 pg/ml for interferon α, 1.37 pg/ml for interferon γ, 0.25 pg/ml for IL-1β, 0.38 pg/ml for IL-6, 0.37 pg/ml for IL-8, 0.62 pg/ml for TNFα, and 11.1 pg/ml for TGFβ.
Change from baseline in joint pain | 4, 12 and 24 weeks
  A Visual Analogic Scale (VAS) for pain at the involved joints will be used for this purpose. Each patient will be invited to indicate the severity of pain by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain". Measurement from the starting point (left end) of the scale to the patients' mark will be recorded in centimeters and will be interpreted as the pain severity.
Change from baseline in DAS score | 4, 12 and 24 weeks
  The DAS (Disease Activity Score) provides a score between 0 and 10, a larger number indicating more active disease. The disease activity is considered ''high"' if DAS is > 5,1, which would mean a worse outcome for the patient's global health; ''moderate" if DAS is > 3,2; ''low'' if DAS is < 3,2; ''on remission'' if DAS is < 2,6, which means a better outcome overall.
Change from baseline in HAQ score | 4, 12 and 24 weeks
  HAQ (Health Assessment Questionnaire) is a quantitative tool used to assess health related quality of life assessments related to many types of injuries or illnesses. Each item or question is rated on a scale of 0 to 3, with 0 (normal/no difficulty), 1 (some difficulty), 2 (much difficulty), and 3 (unable to do). The categories scores are averaged, which represent an overall score from 0 (no disability) to 3 (completely disabled).
Change from baseline in WOMAC index | 4, 12 and 24 weeks
  The Western Ontario and McMaster Universities Arthritis Index (WOMAC) is widely used in the evaluation of Hip and Knee Osteoarthritis. The test questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4).
Change from baseline in CD3, CD8, CD20 at synovial level | 12 weeks
  Similarly for the primary outcome, the analysis of 6 images from each biopsy section will be analysed and the score will be expressed as the mean area of tissue occupied by positively stained cells for each surface protein.
To identify subsets of the disease that could have a better response to the treatment | baseline - 24 weeks
  Two subsets of CPPD have been considered for this study: acute arthritis and chronic CPP crystal inflammatory arthritis. For each subset the changes of clinical, ultrasonographic and patient repoerted outcomes scores will be monitored and compared in order to identify any differences between the the groups. Details on the assessment of such outcomes have been provided above.
To determine changes at ultrasound examination in terms of inflammation and degenerative changes | 4, 12 and 24 weeks
  The ultrasound assessment will include the wrists and hands, knees and the affected joints if different than hands/wrists/knees. Inflammatory changes (synovitis) will be scored according to the semiquantitative Global OMERACT EULAR Scoring System (GLOESS) a semiquantitative score (0-3) that can be interpreted as: no inflammation (0), slight inflammation (1), moderate inflammation (2) and severe inflammation (3) while bone profile irregularities intended as erosions and/or /osteo-proliferative changes (osteophytes) will be scored with a dichotomic score (0: absence, 1:presence). Each site will be scored separately for both inflammatory and bony changes.

OTHER OUTCOMES:
To explore the possible baricitinib-induced impact on whole-body metabolism | 24 weeks
  Untargeted metabolomics analysis on the same samples will be performed using standardized bioinformatics tools to discover the most relevant metabolic pathways involved in the pathogenesis of CPPD and/or valuable to monitor the therapeutic path of the CPPD patient. Targeted metabolomics will be done to quantify key small molecules involved in the energy cycles and oxidative stress. In this analysis, the metabolites will be extracted from the serum and then their concentrations will be compared to the analytical standards.

CONTACTS AND LOCATIONS:
Overall Officials: Georgios Filippou, Assistant Professor, Principal Investigator — IRCCS Galeazzi - Sant&amp;amp;amp;#39;Ambrogio Hospital
Locations (1):
- IRCCS Galeazzi - Sant Ambrogio Hospital, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Krenn V, Morawietz L, Burmester GR, Kinne RW, Mueller-Ladner U, Muller B, Haupl T. Synovitis score: discrimination between chronic low-grade and high-grade synovitis. Histopathology. 2006 Oct;49(4):358-64. doi: 10.1111/j.1365-2559.2006.02508.x. PMID 16978198
- [Background] Krenn V, Morawietz L, Haupl T, Neidel J, Petersen I, Konig A. Grading of chronic synovitis--a histopathological grading system for molecular and diagnostic pathology. Pathol Res Pract. 2002;198(5):317-25. doi: 10.1078/0344-0338-5710261. PMID 12092767
- [Background] Kelly S, Humby F, Filer A, Ng N, Di Cicco M, Hands RE, Rocher V, Bombardieri M, D'Agostino MA, McInnes IB, Buckley CD, Taylor PC, Pitzalis C. Ultrasound-guided synovial biopsy: a safe, well-tolerated and reliable technique for obtaining high-quality synovial tissue from both large and small joints in early arthritis patients. Ann Rheum Dis. 2015 Mar;74(3):611-7. doi: 10.1136/annrheumdis-2013-204603. Epub 2013 Dec 13. PMID 24336336
- [Background] Sirotti S, Terslev L, Filippucci E, Iagnocco A, Moller I, Naredo E, Vreju FA, Adinolfi A, Becce F, Hammer HB, Cazenave T, Cipolletta E, Christiansen SN, Delle Sedie A, Diaz M, Figus F, Mandl P, MacCarter D, Mortada MA, Mouterde G, Porta F, Reginato AM, Schmidt WA, Serban T, Wakefield RJ, Zufferey P, Sarzi-Puttini P, Zanetti A, Damiani A, Pineda C, Keen HI, D'Agostino MA, Filippou G; OMERACT Ultrasound working group-CPPD subgroup. Development and validation of an OMERACT ultrasound scoring system for the extent of calcium pyrophosphate crystal deposition at the joint level and patient level. Lancet Rheumatol. 2023 Aug;5(8):e474-e482. doi: 10.1016/S2665-9913(23)00136-4. Epub 2023 Jul 5. PMID 38251579
- [Background] Terslev L, Naredo E, Aegerter P, Wakefield RJ, Backhaus M, Balint P, Bruyn GAW, Iagnocco A, Jousse-Joulin S, Schmidt WA, Szkudlarek M, Conaghan PG, Filippucci E, D'Agostino MA. Scoring ultrasound synovitis in rheumatoid arthritis: a EULAR-OMERACT ultrasound taskforce-Part 2: reliability and application to multiple joints of a standardised consensus-based scoring system. RMD Open. 2017 Jul 11;3(1):e000427. doi: 10.1136/rmdopen-2016-000427. eCollection 2017. PMID 28948984
- [Background] Uson J, Rodriguez-Garcia SC, Castellanos-Moreira R, O'Neill TW, Doherty M, Boesen M, Pandit H, Moller Parera I, Vardanyan V, Terslev L, Kampen WU, D'Agostino MA, Berenbaum F, Nikiphorou E, Pitsillidou IA, de la Torre-Aboki J, Carmona L, Naredo E. EULAR recommendations for intra-articular therapies. Ann Rheum Dis. 2021 Oct;80(10):1299-1305. doi: 10.1136/annrheumdis-2021-220266. Epub 2021 May 25. PMID 34035002
- [Background] Genovese MC, Smolen JS, Takeuchi T, Burmester G, Brinker D, Rooney TP, Zhong J, Daojun M, Saifan C, Cardoso A, Issa M, Wu WS, Winthrop KL. Safety profile of baricitinib for the treatment of rheumatoid arthritis over a median of 3 years of treatment: an updated integrated safety analysis. Lancet Rheumatol. 2020 Jun;2(6):e347-e357. doi: 10.1016/S2665-9913(20)30032-1. PMID 38273598
- [Background] Caporali R, Taylor PC, Aletaha D, Sanmarti R, Takeuchi T, Mo D, Haladyj E, Bello N, Zaremba-Pechmann L, Fang Y, Dougados M. Efficacy of baricitinib in patients with moderate-to-severe rheumatoid arthritis up to 6.5 years of treatment: results of a long-term study. Rheumatology (Oxford). 2024 Oct 1;63(10):2799-2809. doi: 10.1093/rheumatology/keae012. PMID 38258434
- [Background] Filippou G, Adinolfi A, Cimmino MA, Scire CA, Carta S, Lorenzini S, Santoro P, Sconfienza LM, Bertoldi I, Picerno V, Di Sabatino V, Ferrata P, Galeazzi M, Frediani B. Diagnostic accuracy of ultrasound, conventional radiography and synovial fluid analysis in the diagnosis of calcium pyrophosphate dihydrate crystal deposition disease. Clin Exp Rheumatol. 2016 Mar-Apr;34(2):254-60. Epub 2016 Feb 9. PMID 26886247
- [Background] Abhishek A, Tedeschi SK, Pascart T, Latourte A, Dalbeth N, Neogi T, Fuller A, Rosenthal A, Becce F, Bardin T, Ea HK, Filippou G, Fitzgerald J, Iagnocco A, Liote F, McCarthy GM, Ramonda R, Richette P, Sivera F, Andres M, Cipolletta E, Doherty M, Pascual E, Perez-Ruiz F, So A, Jansen TL, Kohler MJ, Stamp LK, Yinh J, Adinolfi A, Arad U, Aung T, Benillouche E, Bortoluzzi A, Dau J, Maningding E, Fang MA, Figus FA, Filippucci E, Haslett J, Janssen M, Kaldas M, Kimoto M, Leamy K, Navarro GM, Sarzi-Puttini P, Scire C, Silvagni E, Sirotti S, Stack JR, Truong L, Xie C, Yokose C, Hendry AM, Terkeltaub R, Taylor WJ, Choi HK. The 2023 ACR/EULAR classification criteria for calcium pyrophosphate deposition disease. Ann Rheum Dis. 2023 Oct;82(10):1248-1257. doi: 10.1136/ard-2023-224575. Epub 2023 Jul 26. PMID 37495237
- [Background] Tedeschi SK, Huang W, Yoshida K, Solomon DH. Risk of cardiovascular events in patients having had acute calcium pyrophosphate crystal arthritis. Ann Rheum Dis. 2022 Aug 11;81(9):1323-1329. doi: 10.1136/annrheumdis-2022-222387. PMID 35613842
- [Background] Kwan A, Ingrid E, Jiang M, Lim KKT. The cardiovascular risk of JAK inhibitors in treating rheumatic diseases. Int J Rheum Dis. 2024 Aug;27(8):e15308. doi: 10.1111/1756-185X.15308. No abstract available. PMID 39187987
- [Background] Ytterberg SR, Bhatt DL, Mikuls TR, Koch GG, Fleischmann R, Rivas JL, Germino R, Menon S, Sun Y, Wang C, Shapiro AB, Kanik KS, Connell CA; ORAL Surveillance Investigators. Cardiovascular and Cancer Risk with Tofacitinib in Rheumatoid Arthritis. N Engl J Med. 2022 Jan 27;386(4):316-326. doi: 10.1056/NEJMoa2109927. PMID 35081280
- [Background] Damart J, Filippou G, Andres M, Cipolletta E, Sirotti S, Carboni D, Filippucci E, Diez P, Abhishek A, Latourte A, Ea HK, Ottaviani S, Letarouilly JG, Desbarbieux R, Graf S, Norberciak L, Richette P, Pascart T. Retention, safety and efficacy of off-label conventional treatments and biologics for chronic calcium pyrophosphate crystal inflammatory arthritis. Rheumatology (Oxford). 2024 Feb 1;63(2):446-455. doi: 10.1093/rheumatology/kead228. PMID 37216917
- [Background] Zhang W, Doherty M, Pascual E, Barskova V, Guerne PA, Jansen TL, Leeb BF, Perez-Ruiz F, Pimentao J, Punzi L, Richette P, Sivera F, Uhlig T, Watt I, Bardin T. EULAR recommendations for calcium pyrophosphate deposition. Part II: management. Ann Rheum Dis. 2011 Apr;70(4):571-5. doi: 10.1136/ard.2010.139360. Epub 2011 Jan 20. PMID 21257614
- [Background] T Virtanen A, Haikarainen T, Raivola J, Silvennoinen O. Selective JAKinibs: Prospects in Inflammatory and Autoimmune Diseases. BioDrugs. 2019 Feb;33(1):15-32. doi: 10.1007/s40259-019-00333-w. PMID 30701418
- [Background] Guerne PA, Terkeltaub R, Zuraw B, Lotz M. Inflammatory microcrystals stimulate interleukin-6 production and secretion by human monocytes and synoviocytes. Arthritis Rheum. 1989 Nov;32(11):1443-52. doi: 10.1002/anr.1780321114. PMID 2554932
- [Background] Punzi L, Oliviero F, Ramonda R. Transforming growth factor-beta levels in synovial fluid of osteoarthritis with or without calcium pyrophosphate dihydrate crystals. J Rheumatol. 2003 Feb;30(2):420; author reply 420-1. No abstract available. PMID 12583352
- [Background] Martinon F, Petrilli V, Mayor A, Tardivel A, Tschopp J. Gout-associated uric acid crystals activate the NALP3 inflammasome. Nature. 2006 Mar 9;440(7081):237-41. doi: 10.1038/nature04516. Epub 2006 Jan 11. PMID 16407889